CLINICAL TRIAL: NCT02470663
Title: Bone Density in Children With IBD Treated With Amorphous Calcium or Commercial Crystalline Calcium: A Prospective Randomized Multicenter Trial
Brief Title: Bone Density in Children With IBD Treated With Amorphous Calcium or Commercial Crystalline Calcium
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: company and Sheba did not reach an agreement
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Batia Weiss, Director, Pediatric Gastroenterology and Nutrition Unit, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1957-15
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study group (Experimental): Children recieving DENSITYTM caplets (marketed as Amorphical) 200 mg BID for 12 months
  Interventions: Dietary Supplement: DENSITYTM caplets (marketed as Amorphical)
- Control group (Active Comparator): Children recieving Calcium carbonate 600 mg once daily for 12 months
  Interventions: Dietary Supplement: Calcium carbonate 600 mg once daily

INTERVENTIONS:
Dietary Supplement: DENSITYTM caplets (marketed as Amorphical) — supplementation
  Arms: Study group
Dietary Supplement: Calcium carbonate 600 mg once daily — supplementation
  Arms: Control group

SUMMARY:
Patients diagnosed with, or in risk of osteoporosis regularly take calcium dietary supplements, although their contribution to BMD maintenance, prevention of bone loss or reduction of the risk of fracture is questionable. Freshwater crayfish rely on amorphous calcium carbonate (ACC), a thermodynamically instable and very rare biomineralized polymorph of calcium carbonate, as the main mineral in the exoskeleton and in their temporary storage organ, the gastrolith. The study hypothesis is that amorphous calcium carbonate (ACC) will have an advantage over calcium carbonate in improving BMD of pediatric IBD patients with reduced BMD. The investigators will include children 10-18 years old with IBD and reduced bone density to recieve regular calcium or amorphic calcium for 12 months with follow up of bone density and confounders as disease activity and medications.

DETAILED DESCRIPTION:
Abstract- Scientific Background Inflammatory bowel diseases (IBD), including Crohn's disease (CD) and ulcerative Colitis (UC) are chronic disorders of the gastrointestinal tract defined by relapsing and remitting episodes. One of the concerning comorbidities of IBD is reduced bone mineral density (BMD). Recent studies have reported that 43%-46% of children with CD had BMD z-scores <_1 SD at diagnosis (1.2) and that BMD did not improve during treatment for IBD. Chronic inflammation has an adverse effect on skeletal muscle health in children with IBD by multiple mechanisms. Emerging data suggests an increased risk of vertebral fractures in these patients (3). In longitudinal studies, Children with IBD had significantly lower mean BMD z scores for the lumbar spine (LS) at baseline and after 2 years. The reduction occurred in UC and CD, and neither improved their z score during follow-up (4).

Patients diagnosed with, or in risk of osteoporosis regularly take calcium dietary supplements, although their contribution to BMD maintenance, prevention of bone loss or reduction of the risk of fracture is questionable. Freshwater crayfish rely on amorphous calcium carbonate (ACC), a thermodynamically instable and very rare biomineralized polymorph of calcium carbonate, as the main mineral in the exoskeleton and in their temporary storage organ, the gastrolith. Preclinical studies revealed an increase in calcium gastrointestinal bioavailability, bone absorption and retention in rats administered with ACC compared to other calcium supplementation. ACC's beneficial effects on bone loss prevention, bone formation and bone mechanical strength maintenance, was also demonstrated in an ovaryectomy rat model. A clinical study conducted by on 13 postmenopausal women revealed a 2 fold increase in calcium gastrointestinal bioavailability from ACC compared with Calcium Carbonate (5,6). α-Klotho (klotho) is a transmembrane protein which can be cleaved and shed to act as a circulating hormone (7), and is an essential cofactor for the binding of fibroblast growth factor (FGF) to its cognate receptor, serving as a major regulator of phosphate homeostasis (8). Low klotho levels were recently noted in adolescents with anorexia nervosa (9).

Hypothesis

1. Amorphous calcium carbonate (ACC) will have an advantage over calcium carbonate in improving BMD of pediatric IBD patients with reduced BMD.
2. Serum klotho levels will be reduced at the time of IBD diagnosis and will increase following weight rehabilitation. Furthermore, klotho levels will be associated with bone density and with the activity of the GH/IGF-1 axis.

Study Aims

1. To compare the effectiveness of amorphous calcium to calcium carbonate supplementation on MBD improvement in children with IBD and osteopenia/osteoporosis.
2. To compare the tolerability of amorphous calcium to calcium carbonate in children.
3. To assess Klotho levels and their correlation with anthropometric measurements, IGF-I levels, and BMD Z-score, at study entry and completion.

Experimental Design Prospective randomized multicenter investigator blinded trial, including 4 pediatric gastroenterology units.

Study population - Children 10-18 years of age with inflammatory bowel diseases (CD, UC, IBD-U), with proved baseline osteopenia or osteoporosis, measured by lumbar spine Z-score lower than -1.0 (minus 1.0) Inclusion criteria: 1. Children 10-18 years old. 2. Confirmed diagnosis of IBD 3. Able to swallow pills. 4. Osteopenia or osteoporosis (spine Z score lower than -1.0) on baseline bone scan. 5. Informed consent.

Exclusion criteria: 1. Inadequate bone marrow, renal or hepatic function. 2. Significant concurrent disease. 3. Allergy to calcium or vitamin D preparations.

4. Pathologic hypercalciuria. 5. Patient non-compliance. 6. Pregnancy.

Randomization and coding: All sites will be provided with coded numbered opaque envelopes. The envelopes will contain the patient code and randomization to group 1 or group 2. The envelopes must be opened sequentially, and only after informed consent has been obtained. Patients may not be redistributed between treatment arms or reallocated once the envelope is opened. All randomization envelopes will be stored in a safe place and remain unopened until patient is randomized.

Blinding: This is an investigator-blinded study. A pre-packed box with all required medications will be given to the subject after an inform consent is signed. A nurse or physician not involved in the study will address questions and provide further instructions.

Study medication and treatment duration:

Study medication - DENSITYTM caplets (marketed as Amorphical) 200 mg BID. Control medication - Calcium carbonate 600 mg once daily DENSITYTM will be provided by Amorphical company. Vitamin D supplementation - will be given to all patients according to baseline serum level and follow- up, to achieve a sufficient level.

Treatment duration - 52 weeks.

Monitoring -

1. Laboratory tests- Serum calcium, PTH, phosphor, vitamin D - at baseline, and 16, 32, 52 weeks. Urinary calcium (24 hours) - at week 0, 4, 16 and 52 of treatment. Serum and urine bone turnover markers - at baseline and 52 week.
2. Disease activity- by PCDAI, at each visit - every 8-12 weeks
3. Medications records - especially systemic and topical steroid use
4. Diet- dairy product and dietary calcium consumption will be assessed by questionnaires - at baseline, and weeks 16, 32, 52.
5. Compliance - assessed at each visit, by questioning and pill count.
6. Bone mineral density (BMD) - will be performed at baseline and week 52. BMD at the lumbar spine (L1-L4) and the hip will be evaluated using DXA (Lunar Prodigy; GE Medical Systems, Madison, WI, USA). BMD will be expressed in grams per square centimeter and in terms of Z-scores (i.e. the difference between the BMD of the patient and the average BMD of age- and sex-matched controls divided by the standard deviation of the control group). All BMD tests will be performed at Sheba medical center and interpreted by the same physician, who will be blinded to the medication used.
7. Klotho and IGF-1 levels - obtained at baseline and 52 weeks (Samples for klotho and IGF-1 measurements will be centrifuged for 15 minutes at 2700 rpm, separated, and frozen at -70ºC until use. Klotho levels will be analyzed using an α-klotho ELISA kit (Immuno-Biological Laboratories Co, Japan). The kit has been validated and has been widely used for the measurement of klotho levels (10,11).

   IGF-1 will be measured by a chemiluminescent immunometric method (Immulite 2000, Siemens Medical Solutions Diagnostics, Los Angeles, CA, USA).
8. Adverse events- will be followed through week 60.

Primary endpoint The primary efficacy endpoint is improvement of spine bone density by 0.5 points in Z -score after 12 months.

Secondary endpoints

1. Improvement of spine bone density by at least 0.25 points in Z -score after 12 months.

Sample size Sample size was calculated based on the assumption that the primary endpoint will be achieved in 20% of patients on the standard calcium+D, supplementation and in 40% of patients on the study medication.

The sample size is 50 patients in each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Children 10-18 years old.
2. Confirmed diagnosis of IBD
3. Able to swallow pills.
4. Osteopenia or osteoporosis (spine Z score lower than -1.0) on baseline bone scan.
5. Informed consent.

Exclusion Criteria:

1. Inadequate bone marrow, renal or hepatic function.
2. Significant concurrent disease.
3. Allergy to calcium or vitamin D preparations.
4. Pathologic hypercalciuria. 5. Patient non-compliance. 6. Pregnancy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint is improvement of spine bone density by 0.5 points in Z -score after 12 months | 12 months

SECONDARY OUTCOMES:
Improvement of spine bone density by at least 0.25 points in Z -score after 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Batia Weiss, MD, Principal Investigator — Sheba Medical Center

REFERENCES:
- [Background] Schmidt S, Mellstrom D, Norjavaara E, Sundh SV, Saalman R. Low bone mineral density in children and adolescents with inflammatory bowel disease: a population-based study from Western Sweden. Inflamm Bowel Dis. 2009 Dec;15(12):1844-50. doi: 10.1002/ibd.20962. Epub 2009 Apr 30. PMID 19408319
- [Background] Sylvester FA, Wyzga N, Hyams JS, Davis PM, Lerer T, Vance K, Hawker G, Griffiths AM. Natural history of bone metabolism and bone mineral density in children with inflammatory bowel disease. Inflamm Bowel Dis. 2007 Jan;13(1):42-50. doi: 10.1002/ibd.20006. PMID 17206638
- [Background] Schmidt S, Mellstrom D, Norjavaara E, Sundh V, Saalman R. Longitudinal assessment of bone mineral density in children and adolescents with inflammatory bowel disease. J Pediatr Gastroenterol Nutr. 2012 Nov;55(5):511-8. doi: 10.1097/MPG.0b013e31825817a0. PMID 22688562
- [Background] Wong SC, Catto-Smith AG, Zacharin M. Pathological fractures in paediatric patients with inflammatory bowel disease. Eur J Pediatr. 2014 Feb;173(2):141-51. doi: 10.1007/s00431-013-2174-5. Epub 2013 Oct 17. PMID 24132387
- [Result] Shaltiel, G., Bar-David, E., Meiron, O. E., et al. Bone loss prevention in ovariectomized rats using stable amorphous calcium carbonate. Health 2013; 5 (7A2): 18-29
- [Result] Vaisman N, Shaltiel G, Daniely M, Meiron OE, Shechter A, Abrams SA, Niv E, Shapira Y, Sagi A. Increased calcium absorption from synthetic stable amorphous calcium carbonate: double-blind randomized crossover clinical trial in postmenopausal women. J Bone Miner Res. 2014 Oct;29(10):2203-9. doi: 10.1002/jbmr.2255. PMID 24753014